CLINICAL TRIAL: NCT02752893
Title: Estrogen Receptor-Positive Breast Cancer Patient-Derived Xenografts
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Gary Schwartz, Staff Physician, Hematology-Oncology, Dartmouth-Hitchcock Medical Center
Other Study IDs: D16100
Record Dates: First submitted 2016-04-26; First posted 2016-04-27 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
Keywords: estrogen; estrogen receptor; ER+; HER2; HER2-; HER2-negative; xenograft; co-clinical; mice; patient-derived xenograft; patient-derived; breast cancer; precision medicine; personalized medicine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators will establish a platform at Dartmouth-Hitchcock Medical Center to generate novel models of estrogen receptor alpha-positive (ER+), human epidermal growth factor receptor 2-negative (HER2-) breast cancer, which will be used for research studies to develop novel treatment strategies and dissect signaling pathways underlying drug sensitivity and resistance.

ELIGIBILITY:
Inclusion criteria

1. Men and women > age 18 with histologically documented ER+/HER2- breast cancer or with a history of ER+/HER2- breast cancer, for whom a tumor biopsy or surgical resection is clinically indicated and will be performed as standard of care.

   Tumor specimens may be from breast (progressive or recurrent) or metastatic sites. Patients with multicentric or bilateral disease are eligible.
2. Patients must have disease progression during neoadjuvant therapy, recurrence after neoadjuvant or adjuvant therapy, or progression after systemic therapy for metastatic disease.
3. ER positivity is defined as >10% of malignant tumor cells staining positively for ER by immunohistochemistry (IHC).

   HER2 negativity is defined as IHC 0-1+, or with a fluorescence in situ hybridization (FISH) ratio of <1.8 if IHC is 2+ or if IHC has not been done.
4. Excess LIVE tumor tissue must be available from the surgically resected tumor specimen, or from 1-3 extra core needle or incisional biopsy. LIVE tumor tissue must be available within 2 hours of removal from patient (shorter time is preferable).
5. A recurrent or progressing breast cancer must be greater than 1 cm in greatest diameter.
6. Prior therapy is allowed as long as excess viable tumor tissue is available from the biopsy or surgical excision procedure.
7. Patients must be willing to provide 6 mL of blood, which can be obtained during a routine clinically indicated blood draw (ideally, done on the same day as the tumor biopsy/surgery).
8. Ability to give signed informed consent.

Exclusion Criteria

1. Fine needle aspirates and effusions of bodily fluids are not eligible as sources of tumor cells.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects >18 years of age with disease progression during neoadjuvant therapy, recurrence after neoadjuvant or adjuvant therapy, or progression after systemic therapy for metastatic disease that expresses estrogen receptor alpha (ER+) and does not overexpress HER2 (HER2-, HER2-negative).
  Subjects must be scheduled to undergo a clinically indicated biopsy or surgical removal of tumor, and excess tumor tissue must be available for research use.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Xenograft success rate, defined as the percentage of patient tumors that yield a growing xenograft in mice. | 1 year from time of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No